

H-4032 Debrecen, Nagyerdei krt. 98. Tel/fax: 52/411-717/56732, email: fokdh@dental.unideb.hu

| Identification number: | Code: |
|------------------------|-------|

# **Informed Consent**

## Place of the study:

University of Debrecen, Clinical Center, Faculty of Dentistry

#### **Address and contact:**

Address: 4032, Debrecen, Nagyerdei körút 98.

Phone number: +36 52 255 208

Correspondence: 4002 Debrecen, Pf. 400., UD, Faculty of Dentistry

## Name of the study director:

Dr. Kinga Ágnes Bágyi (Dean, associate professor)

#### Personal data:

- Name:
- Date of birth:
- Health insurance:
- Mother's name:
- Address:
- Contact:

**Supplement 2: Informed consent - Effect of Sour Cherry Anthocyanins on Human Salivary Cariogenic Biofilm Formation** 

#### KLINIKAI KÖZPONT FOGORVOSI SZOLGÁLAT



H-4032 Debrecen, Nagyerdei krt. 98. Tel/fax: 52/411-717/56732, email: fokdh@dental.unideb.hu

| Undersigned, |
|---|
| I declare, that I could ask about the study and I got answer to my questions about the study. I got answer to my every questions. I understand the conditions and I accept them. |
| I agree with the participation in the study and I voluntarily participaate in the experiment. |
| I know that I don't get any allowance for the participation. |
| I understand that I can cancel my participation at any time during the study. I contribute with my signature to use my personal data, involving data about my physical or spiritual health, my ancestry and sample materials are used as it was mentioned during the information with an identification number instead of my name. |
| I know that I will get one copy from this Informed consent paper. |
| signature |
| Debrecen, |
| signature of the participant |
| The name and workplace status of the doctor who gave the information: |